CLINICAL TRIAL: NCT06370507
Title: Ventilation Monitoring by Electrical Impedance Tomography During Anesthesia for Pediatric Surgery: an Observational Prospective Data-registry
Brief Title: Monitoring of Lung Ventilation Through Electrical Impedance Tomography During Pediatric Surgery
Acronym: VentiPed
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Gianmaria Cammarota, MD, PhD, Associate Professor, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Other Study IDs: UPO2#
Record Dates: First submitted 2024-04-06; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Ventilator Lung; Surgery; Pediatric
Keywords: Electrical impedance tomography; Surgery; Pediatric
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients undergoing sedation or general anesthesia: Pediatric patients undergoing sedation or general anesthesia subjected to ventilation distribution assessment via electrical impedance tomography
  Interventions: Device: Electrical impedance tomography assessment of ventilation distribution in course of sedation/general anesthesia for pediatric surgery

INTERVENTIONS:
Device: Electrical impedance tomography assessment of ventilation distribution in course of sedation/general anesthesia for pediatric surgery — Assessment of ventilation distribution through electrical impedance tomography in pediatric patients subjected to sedation or general anesthesia for surgery

SUMMARY:
Given the scarcity of studies aimed at assessing the effect of anesthesia and m ventilation on the distribution of lung ventilation in pediatric patients undergoing surgery, with the exclusion of thoracic surgery, the present prospective observational study would shed the light on ventilation practice in pediatric anesthesia for surgery. This study wold fill the actual gap allowing the evaluation, through electrical impedance tomography (EIT) of the distribution of lung ventilation across the different phases of anesthesia for pediatric surgery. These insights could contribute to improve clinical practice and research in the management of ventilation in pediatric patients undergoing anesthesia for surgery.

DETAILED DESCRIPTION:
Anesthesia for surgery is associated with the development of atelectasis and hypoventilation that may persist postoperatively, exposing patients to postoperative pulmonary complications. The main cause is the loss of muscle tone, especially of the diaphragm, which is affected by the pressure exerted by the abdominal viscera, resulting in elevation and compression of alveoli and small airways in the posterior lung regions, leading to collapse and atelectasis, as well as redistribution of ventilation. These variations are even more pronounced in pediatric patients, who have significantly greater chest wall compliance and markedly lower functional residual capacity compared to adults, making them physiologically predisposed to derecruitment during anesthesia. These phenomena are well recognized, but their magnitude and causes are relatively poorly documented due to the scarcity of means capable of precise assessment. EIT is an extremely useful tool as it allows real-time monitoring of changes in the topographic distribution of ventilation in a completely non-invasive manner, highlighting atelectasis and redistribution of aeration. EIT is an imaging technique used in both pediatric and adult patients, analyzing tissue resistivity properties against low-intensity currents applied to the chest via electrodes placed at the IV-VI intercostal spaces. Scans are generated from the collected potential differences and known excitation currents using weighted back-projection into a matrix of pixels. Each pixel represents the instantaneous relative local impedance change compared to a baseline, caused by the presence of a larger or smaller volume of air. This allows for real-time and precise reconstruction of lung air distribution for each breath using dedicated software. In adults, its application in the operating room allows monitoring of lung ventilation distribution during anesthesia, mechanical ventilation, and surgical procedures capable of altering it (such as pneumoperitoneum), optimizing ventilatory settings to avoid atelectasis and derecruitment. Studies in the pediatric field have shown great promise but are significantly limited, mostly conducted in extreme age groups (premature and neonatal) and almost exclusively during spontaneous breathing and without sedation. Pediatric patients undergo a series of respiratory system modifications from birth to adolescence due to lung and alveolar growth, ossification of the rib cage, and muscle tone increase, making the generalization of parameters and findings impossible. Children undergo a series of respiratory system modifications from birth to adolescence due to lung and alveolar growth, ossification of the rib cage, and increased muscle tone, making it impossible to generalize physiological parameters and findings that can vary significantly across different age groups (neonate, infant, preschool-age child, child, adolescent).

Given the scarcity of studies aimed at assessing the effect of anesthesia and surgical technique on the distribution of lung ventilation in pediatric patients undergoing surgery, with the exclusion of thoracic surgery, the present prospective observational study would shed the light on ventilation practice in pediatric anesthesia for surgery. This study wold fill the actual gap allowing the evaluation, through EIT of the distribution of lung ventilation across the different phases of anesthesia for pediatric surgery. These insights could contribute to improve clinical practice and research in the management of ventilation in pediatric patients undergoing anesthesia for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents under 14 years of age
2. Elective and urgent surgeries, excluding thoracic surgeries, managed with any anesthesia modality, including:

   * Deep sedation with spontaneous breathing associated with regional anesthesia
   * Deep sedation with the use of a laryngeal mask for airway control and ventilatory support
   * General anesthesia with endotracheal tube placement
   * American Society of Anesthesiologists (ASA) I-III classification
   * Negative medical history for airway infection with fever in the two weeks preceding the study, three weeks for patients with a personal history of laryngospasm and bronchospasm.

Exclusion Criteria:

* Age > 14 years
* ASA > III
* Known lung pathology
* Lack of parental consent for the study
* Occurrence of serious complications during anesthesia (such as laryngospasm or bronchospasm)

Ages: 0 Days to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents under the age of 14 who need to undergo surgical procedures excluding thoracic surgery.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Ventilation distribution | Intraoperative time frame
  Ventilation distribution assessment through Electrical impedance tomography

SECONDARY OUTCOMES:
Intraoperative ventilatory respiratory mechanics | Intraoperative time frame
  Respiratory mechanics
Postoperative pulmonary complications | Immediately after surgery till 7th day after intervention or hospital discharge
  Postoperative pulmonary complications (pneumonia, acute respiratory distress syndrome, atelectasis requiring supplemental oxygen administration or non-invasive respiratory support or invasive mechanical ventilation)
Intraoperative oxygenation | Intraoperative time frame
  Oxygenation evaluated through peripheral oxygen saturation
Intraoperative hemodynamics | Intraoperative time frame
  blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Gianmaria Cammarota, Prof, Principal Investigator — Università degli Studi del Piemonte Orientale Amedeo Avogadro

REFERENCES:
- [Derived] Rosalba D, Meneghetti G, Verdina F, Solai C, Azzolina D, Petronio L, Guaraglia M, Buscaglia R, Saviolo G, Furlan G, Vietti F, Biasucci D, Spadaro S, Simonte R, De Robertis E, Longhini F, Penpa S, Ubertazzi M, Panuccio E, Aluffi P, De Cilla S, Brucoli M, Vaschetto R, Cammarota G. Patterns of lung aeration assessed through electrical impedance tomography in paediatric patients undergoing elective surgery: insights from a prospective and observational data-registry. J Anesth Analg Crit Care. 2025 Jun 23;5(1):34. doi: 10.1186/s44158-025-00254-x. PMID 40551255